CLINICAL TRIAL: NCT05321654
Title: The Effects of Postural Education or Corrective Exercise Intervention on the Craniovertebral Angle in Young Adults With Forward Head Posture: A Randomized Controlled Trial
Brief Title: Effects of Postural Education or Corrective Exercise on Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberty University (Other)
Collaborators: National Academy of Sports Medicine (Unknown)
Responsible Party: Principal Investigator, Dr. David Titcomb, Professor of Health Sciences, Liberty University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY20-21-1073; UR2201 (Other Grant/Funding Number: Liberty University Center for Research & Scholarship)
Record Dates: First submitted 2022-03-18; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Postural; Defect
Keywords: Forward Head Posture; Craniovertebral Angle; Corrective Exercise Program; Postural Education
MeSH Terms: interventions — Educational Status; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: A prospective parallel randomized controlled trial with repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Posture Education (PE) Group (Experimental): PE group members received a 20-minute in-person one-on-one standardized educational session by a research team member in the laboratory on the following topics: health risks associated with forward head posture; postural guidelines for using mobile electronic devices, desktop computers, and laptop computers; as well as rest break guidelines. Participants were asked to adhere to the postural guidelines provided in the educational session for the next 4 weeks.
  Interventions: Behavioral: Education for Behavior Modification
- Self-Myofascial Release + Stretching (SMRS) Group (Experimental): This group applied self-myofascial release (SMR) to their thoracic spine with a myofascial roller for 30 sec., then 6 repetitions of myofascial rolling for 90 sec. They applied SMR for 30 sec. to their neck flexors and extensors using their fingertips. They applied SMR to the upper trapezius and pectoralis for 30 sec using a soft tissue mobilization tool. For the first 2 weeks, they performed SMR 3x/wk. During wks. 3 and 4, they progressed SMR to 5 days/wk. Group members also performed stretching to these same muscles after SMR 3 days/wk for the first 2 weeks of the study, progressing to 5 days/wk during weeks 3 and 4.
  Interventions: Behavioral: Corrective Exercise Program
- Self-Myofascial Release + Stretching + Strengthening (SMRSS) Group (Experimental): This group performed the same protocol as SMRS group, as well as include the following strengthening exercises: the supine chin tuck (SCT), upper thoracic-lower cervical extension (UTLCE) using an exercise band that provided 5.5 pounds of resistance, and a single-arm row with trunk rotation (SARTR) using exercise tubing that provided 20 pounds of resistance. The SCT was progressed in 3 phases: Week 1: chin tuck held 2 sec., 5 reps. Week 2: same as week 1, but included us of a towel roll placed under the head. Wks. 3 and 4: chin tuck with head lift 1 in., 2 sec. hold. UTLCE: neck extension with exercise band, held 2 sec. SARTR: single arm row with trunk rotation was performed in a controlled and fluid manner using a self-selected speed. The UTLCE and SARTR were performed with 1 X 10 reps for wks 1-2 and progressed to 2 X10 reps in wks 3-4. Strengthening exercises were performed 3x/wk. for 4 wks.
  Interventions: Behavioral: Corrective Exercise Program
- Control Group (CG) (No Intervention): Participants in the CG did not receive an intervention.

INTERVENTIONS:
Behavioral: Education for Behavior Modification — Please see arm description for a detailed description of the intervention
  Arms: Posture Education (PE) Group
Behavioral: Corrective Exercise Program — Please see arm description for a detailed description of the intervention
  Arms: Self-Myofascial Release + Stretching (SMRS) Group; Self-Myofascial Release + Stretching + Strengthening (SMRSS) Group

SUMMARY:
This randomized control trial examined the effects of postural education or corrective exercise intervention on the craniovertebral angle (CVA) in young adults with forward head posture (FHP). The objectives were 1: to investigate whether or not a corrective exercise program (CEP) consisting of self-myofascial release (SMR) + stretching; a CEP consisting of SMR + stretching + strengthening; or postural education (PE) had an effect on the CVA; 2. to determine which intervention yielded the greatest postural enhancement if a positive effect was observed in more than one intervention. *[note: SMR is a technique involving the self-application of pressure to fascia and muscle tissue for the purpose of enhancing flexibility, reducing muscle soreness, and influencing muscle relaxation]. It was hypothesized that 4 weeks after receiving either CEP intervention or PE there would be a significant change in the CVA compared to a control group; and that there would be an intervention more effective than the others for improving the CVA. The null hypotheses were: there would be no CVA change after intervention in any of the groups; and there will be no intervention more effective than another for improving the CVA.

DETAILED DESCRIPTION:
A total of 94 participants responded to invitations to voluntarily participate and completed the Physical Activity Readiness Questionnaire (PAR-Q+), followed by a questionnaire to rate their current stage of change (SOC) from the Transtheoretical Model adapted to assess exercise/postural modification behavior change (this will be discussed further in eligibility section). On this questionnaire, participants also responded to a yes/no question regarding if they have had a recent injury to their head, shoulders, or spine; or have ever been diagnosed with a pathology related to their cervical/thoracic spine or extremities, as part of exclusion criteria for the study. Participants then underwent a head posture screening performed by the primary investigator who is a licensed physical therapist in the Liberty University Biomechanics & Motion Analysis Laboratory with the use of photogrammetry (use of a digital camera and software to measure posture) as described below.

Participants were asked to arrive at the lab wearing either a tank top or t-shirt, as well as to have their hair tied back if necessary. Height and weight were measured using a digital scale (Health-o-meter Professional, model 500KL, McCook, IL). Participants were instructed to sit comfortably on a stool with hands resting approximately two-thirds down their thighs with palms supinated and feet flat on the ground with hips and knees at 90 degrees; and to look straight ahead at an opposite wall in the laboratory. A digital camera (Canon Powershot, model SX540, Tokyo, Japan) was mounted and leveled on a tripod (Manfrotto, model 055, Cassola, IT) and placed three meters away from the subject. Two photographs were taken of participant's posture. Immediately after data capture, image files were uploaded into Kinovea video analysis software (version 8.15) for CVA assessment. CVA assessment will be discussed further in outcome measures section.

Seventy-nine participants met inclusion criteria (discussed in detail in future section) and were enrolled in the study. Randomization of participant group assignments was completed by the PI using a block randomization generator. Utilizing a sequence created by the block randomizer, the PI placed participants who met inclusion criteria into one of four groups: postural education (PE; n = 20), self-myofascial release + stretching (SMRS; n = 20), self-myofascial release + stretching + strengthening (SMRSS; n = 19), and control group (CG; n = 20). Details of these groups will be provided in future sections. A hard-copy of the sequence generator report was kept concealed in a manila folder and was only opened by the PI during group delegation.

Intervention duration was 4 weeks. Two weeks into the study, participants in intervention groups completed a mid-study questionnaire to assess intervention compliance. At the end of the study (after the completion of 4 weeks) participants in intervention groups completed a post-study questionnaire to assess intervention compliance. All study participants were asked to return back to the Biomechanics laboratory after the completion of the 4 week intervention period to undergo follow-up posture screening, which followed the same posture assessment procedures as described above.

Declarations of interest: This study was part of the requirements for completion of a Ph.D. dissertation (Concordia University Chicago) by David Titcomb, DPT.

Conflicts of interest: none.

ELIGIBILITY:
Inclusion Criteria:

* Completion of informed consent
* Craniovertebral angle ≤ 53 degrees
* Self-rating of Transtheoretical Model stage of change stage ≥ 3/5

Exclusion Criteria:

* Any musculoskeletal injury to the head, shoulders, or spine within the last six months
* Diagnosis of pathology related to the cervical spine, thoracic spine, or upper extremities
* Non-clearance for physical activity based on results of the 2020 PAR-Q+ questionnaire

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Change in Craniovertebral Angle after 4 weeks | Baseline: On day 1 of study enrollment; Post-Intervention: Within 5 days after the end of the 4 week intervention period
  The angle between the intersection of two lines drawn on the photograph: the first line drawn from the tragus of the ear to the spinous process of C7 vertebrae and the second line drawn horizontally through C7 spinous process. In this study, a second researcher directly observed the primary investigator performing each CVA assessment, as well as provided verbal agreement with the accuracy of angle measurement. For each participant, the CVA was derived by taking the mean of two CVA measurements that were assessed on the captured photographs.

SECONDARY OUTCOMES:
Midpoint Intervention Compliance | Assessed at the start of week 3
  On a questionnaire, participants were asked to rate their compliance with their assigned intervention guidelines. Consistent. 75% adherence to guidelines; Moderately Consistent. 50 to 75% adherence to guidelines; Inconsistent. Less than 50% adherence to guidelines.
Endpoint Intervention Compliance | Within 5 days after the end of the 4 week intervention period.
  On a questionnaire, participants were asked to rate their compliance with their assigned intervention guidelines. Consistent. 75% adherence to guidelines; Moderately Consistent. 50 to 75% adherence to guidelines; Inconsistent. Less than 50% adherence to guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: David A Titcomb, DPT, Principal Investigator — Liberty University; Bridget F Melton, EdD, Study Chair — Concordia University Chicago; Theresa Miyashita, PhD, Study Director — Concordia University Chicago; Helen W Bland, PhD, Study Director — Concordia University Chicago
Locations (1):
- Liberty University, Lynchburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting immediately after publication. No end date.
Access Criteria: The primary investigator will review requests received by email. Requests granted to researchers and/or research institutions for the purpose of future research studies. The Liberty University Institutional Review Board will also be notified prior to releasing IPD and/or supporting information. Rather than a URL, individuals interested in IPD and/or supporting information will contact the primary investigator by email, which will be provided in the publication along with a statement about the plan to share IPD.

REFERENCES:
- [Background] Abdelhameed AA, Abdel-Aziem AA. Exercise training and postural correction improve upper extremity symptoms among touchscreen smartphone users. Hong Kong Physiother J. 2016 Sep 7;35:37-44. doi: 10.1016/j.hkpj.2016.06.001. eCollection 2016 Dec. PMID 30931032
- [Background] Bayattork M, Seidi F, Minoonejad H, McClure P, Mozafaripoor E. Intra-rater and inter-rater reliability and agreement of the scapular dyskinesis test in young men with forward head and round shoulder posture. J Rehabil. Sci. 2019 Dec 10;6(4):169-173. https://doi.org/10.30476/JRSR.2019.82944.1037
- [Background] Carter SE, Draijer R, Holder SM, Brown L, Thijssen DHJ, Hopkins ND. Regular walking breaks prevent the decline in cerebral blood flow associated with prolonged sitting. J Appl Physiol (1985). 2018 Sep 1;125(3):790-798. doi: 10.1152/japplphysiol.00310.2018. Epub 2018 Jun 7. PMID 29878870
- [Background] Cuellar JM, Lanman TH. "Text neck": an epidemic of the modern era of cell phones? Spine J. 2017 Jun;17(6):901-902. doi: 10.1016/j.spinee.2017.03.009. Epub 2017 Mar 20. No abstract available. PMID 28336483
- [Background] Engelmann C, Schneider M, Kirschbaum C, Grote G, Dingemann J, Schoof S, Ure BM. Effects of intraoperative breaks on mental and somatic operator fatigue: a randomized clinical trial. Surg Endosc. 2011 Apr;25(4):1245-50. doi: 10.1007/s00464-010-1350-1. Epub 2010 Sep 11. PMID 20835716
- [Background] Fahmy R. NASM Essentials of corrective exercise training. 2nd ed. Burlington, Massachusetts: Jones & Bartlett Learning; 2022.
- [Background] Gustafsson E. Ergonomic recommendations when texting on mobile phones. Work. 2012;41 Suppl 1:5705-6. doi: 10.3233/WOR-2012-0925-5705. PMID 22317659
- [Background] Hansraj KK. Assessment of stresses in the cervical spine caused by posture and position of the head. Surg Technol Int. 2014 Nov;25:277-9. PMID 25393825
- [Background] Kalichman L, Bulanov N, Friedman A. Effect of exams period on prevalence of Myofascial Trigger points and head posture in undergraduate students: Repeated measurements study. J Bodyw Mov Ther. 2017 Jan;21(1):11-18. doi: 10.1016/j.jbmt.2016.04.003. Epub 2016 Apr 7. PMID 28167166
- [Background] Kar G, Hedge A. Effect of workstation configuration on musculoskeletal discomfort, productivity, postural risks, and perceived fatigue in a sit-stand-walk intervention for computer-based work. Appl Ergon. 2021 Jan;90:103211. doi: 10.1016/j.apergo.2020.103211. Epub 2020 Aug 17. PMID 32818838
- [Background] Kim BB, Lee JH, Jeong HJ, Cynn HS. Effects of suboccipital release with craniocervical flexion exercise on craniocervical alignment and extrinsic cervical muscle activity in subjects with forward head posture. J Electromyogr Kinesiol. 2016 Oct;30:31-7. doi: 10.1016/j.jelekin.2016.05.007. Epub 2016 May 24. PMID 27261928
- [Background] Kim SY, Koo SJ. Effect of duration of smartphone use on muscle fatigue and pain caused by forward head posture in adults. J Phys Ther Sci. 2016 Jun;28(6):1669-72. doi: 10.1589/jpts.28.1669. Epub 2016 Jun 28. PMID 27390391
- [Background] Kuroda Y, Sato Y, Ishizaka Y, Yamakado M, Yamaguchi N. Exercise motivation, self-efficacy, and enjoyment as indicators of adult exercise behavior among the transtheoretical model stages. Glob Health Promot. 2012 Mar;19(1):14-22. doi: 10.1177/1757975911423073. Epub 2012 Feb 14. PMID 24801311
- [Background] Lau KT, Cheung KY, Chan KB, Chan MH, Lo KY, Chiu TT. Relationships between sagittal postures of thoracic and cervical spine, presence of neck pain, neck pain severity and disability. Man Ther. 2010 Oct;15(5):457-62. doi: 10.1016/j.math.2010.03.009. PMID 20430685
- [Background] Lee DY, Nam CW, Sung YB, Kim K, Lee HY. Changes in rounded shoulder posture and forward head posture according to exercise methods. J Phys Ther Sci. 2017 Oct;29(10):1824-1827. doi: 10.1589/jpts.29.1824. Epub 2017 Oct 21. PMID 29184298
- [Background] Neupane S, Ali UI, Mathew A. Text neck syndrome-systematic review. Imp. J. Interdiscip. Res. 2017; 3(7): 141-148. http://www.onlinejournal.in
- [Background] Richards KV, Beales DJ, Smith AJ, O'Sullivan PB, Straker LM. Neck Posture Clusters and Their Association With Biopsychosocial Factors and Neck Pain in Australian Adolescents. Phys Ther. 2016 Oct;96(10):1576-1587. doi: 10.2522/ptj.20150660. Epub 2016 May 12. PMID 27174256
- [Background] Ruivo RM, Pezarat-Correia P, Carita AI. Cervical and shoulder postural assessment of adolescents between 15 and 17 years old and association with upper quadrant pain. Braz J Phys Ther. 2014 Jul-Aug;18(4):364-71. doi: 10.1590/bjpt-rbf.2014.0027. Epub 2014 Jul 18. PMID 25054381
- [Background] Sahu M, Sundari KG, David A. Recent ergonomic interventions and evaluations on laptop, smartphones and desktop computer users. In Arockiarajan A, Duraiselvam M, Raju R, editors. Advances in Industrial Automation and Smart Manufacturing. Singapore: Springer; 2021. p. 207-224. https://doi.org/10.1007/978-981-15-4739-3
- [Background] Syamala KR, Ailneni RC, Kim JH, Hwang J. Armrests and back support reduced biomechanical loading in the neck and upper extremities during mobile phone use. Appl Ergon. 2018 Nov;73:48-54. doi: 10.1016/j.apergo.2018.06.003. Epub 2018 Jun 18. PMID 30098642
- [Background] Vate-U-Lan P. Text neck epidemic: a growing problem for smart phone users in Thailand. Int J Comput. Internet Manage. 2015 Sept-Dec;23(3): 551-556.
- [Background] Warburton DER, Jamnik VK, Bredin SSD, and Gledhill N. The physical activity readiness questionnaire for everyone (PAR-Q+) and electronic physical activity readiness medical examination (ePARmed-X+). Health Fit J of Canada. 2011; 4(2):3-23. https://doi.org/10.14288/hfjc.v4i2.103

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT05321654/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT05321654/ICF_001.pdf